CLINICAL TRIAL: NCT01809483
Title: Comparison Between Bandage Contact Lens and Pressure Patching for The Erosion Area and Pain Scale in Corneal Erosion Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Ni Nyoman Triharpini, Resident in Depatment of Ophthalmology Faculty of Medicine, Udayana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LB0201/IIC5D11/16095/2012
Record Dates: First submitted 2013-03-08; First posted 2013-03-12 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Erosion; Cornea, Traumatic
Keywords: mechanical corneal erosion; bandage contact lens; pressure patching; erosion area; pain scale
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bandage contact lens group (Experimental): subject received antibiotic eye drops (combination of Polymyxin B, neomycin and gramicidin, q.i.d), and cycloplegic eye drops (tropicamide 0,5 %, q.d) and bandage contact lens. Bandage contact lenses maintained for 24 hours. Antibiotic eye drops were instilled without removing the contact lenses
  Interventions: Device: Bandage contact lens
- Pressure patching group (Active Comparator): Subject received antibiotic eye drops (combination of Polymyxin B, neomycin and gramicidin, q.i.d), and cycloplegic eye drops (tropicamide 0,5 %, q.d) and pressure patching. Pressure patching maintained for 24 hours and only opened for drug application. Subject and their families were educated on how to perform a good pressure patching
  Interventions: Device: Pressure patching

INTERVENTIONS:
Device: Bandage contact lens — Bandage contact lens : contact lenses (material senofilcon A; base curve 8,8 mm; power - 0,50; diameter 14 mm)
  Arms: Bandage contact lens group
Device: Pressure patching — Pressure patching : using 2 pieces of sterile gauze. The first gauze placed vertically and the second placed horizontally, then fixed with adhesive tape so that eyelid can not move.
  Arms: Pressure patching group

SUMMARY:
This research aims to compare between bandage contact lens and pressure patching in reducing size of erosion area and pain scale in corneal erosion patients as well as its complications.

DETAILED DESCRIPTION:
This is a randomized open-label clinical trial in patients with mechanical corneal erosion. Subjects were selected to use bandage contact lens (Senofilcon A) or pressure patching. All subjects received combination of Polymyxin B, Neomycin, and Gramicidin eye drops and 0,5% Tropicamide eye drops. Evaluation was done 24 hours after treatment

ELIGIBILITY:
Inclusion Criteria:

* aged 17-55 years
* onset of corneal erosion < 48 hours
* corneal erosion due to mechanical injury
* extensive corneal erosion > 3 mm2

Exclusion Criteria:

* bilateral corneal erosion
* corneal erosion due to chemical or thermal injury
* history of systemic analgesic use within 1 week prior to the examination or topical analgesics within 1 hour before the examination
* history of systemic or topical antibiotics within 1 week prior to the examination
* other abnormalities due to trauma
* palpebral or eyelashes position abnormalities
* anterior segment infections
* tear break-up time < 7 seconds in the contra lateral eye

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Size of corneal erosion area | 24 hour
  Corneal erosion area is the multiplication of the long and short axis of corneal erosion, as measured using a caliper, with the help of fluorescein and cobalt blue slit lamp beam

SECONDARY OUTCOMES:
Pain scale | 24 hour
  Pain scale assessment conducted using the Visual Analogue Scale (VAS) subjectively

OTHER OUTCOMES:
Complication | 24 hour
  Complication of corneal erosion (e.g. conjunctivitis, keratitis, corneal ulcer)

CONTACTS AND LOCATIONS:
Overall Officials: Ni Nyoman Triharpini, MD, Principal Investigator — Department of Ophthalmology, Medical Faculty Udayana University / Sanglah Public General Hospital
Locations (1):
- Depatment of Ophthalmolohy, Medical Faculty, Udayana University / Sanglah Public General Hospital, Denpasar, Bali, Indonesia